CLINICAL TRIAL: NCT04018612
Title: A Randomized, Double-Blind, Multi-Dose, Single-Site, Placebo- and Active-Controlled, Efficacy, Tolerability, Safety and Pharmacokinetic Study of Two Different Dosing Regimens of Acetaminophen in Post-Surgical Dental Pain.
Brief Title: A Study of Acetaminophen for Post Surgical Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nevakar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-NVK009-0002
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative; Dental Pain
MeSH Terms: conditions — Pain, Postoperative; Toothache | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: High Dose Acetaminophen (APAP) versus Placebo, Low Dose APAP versus Placebo
Who Masked: Participant, Investigator
Masking Description: Double Blind, Placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose Acetaminophen (Active Comparator): High Dose Acetaminophen Post Op
  Interventions: Drug: Acetaminophen
- Low Dose Acetaminophen (Active Comparator): Low Dose Acetaminophen Post Op
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Placebo Post Op
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen is an analgesic and antipyretic
  Other Names: APAP
  Arms: High Dose Acetaminophen; Low Dose Acetaminophen
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
To assess the safety, tolerability, analgesic, efficacy and pharmacokinetics of high dose acetaminophen relative to placebo and low dose acetaminophen relative to placebo over a 24 hour period in patient experiencing moderate to severe pain following the surgical removal of third molar.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, single-site, placebo-controlled, parallel-group study to assess similarities in safety, tolerability, efficacy, and pharmacokinetics of high dose acetaminophen given relative to placebo, and low dose acetaminophen given relative to placebo over a 24-hour period in patients experiencing moderate to severe postsurgical pain within 7 hours following surgical removal of 2 or more molars

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be capable of reading, comprehending, and signing the informed consent/assent form;
2. Male and female patients between 17-55 years of age;
3. Body Mass Index (BMI) ≤35.0 kg/m2
4. Body weight of >50 kg
5. Patients are American Society of Anaesthesiologists (ASA) Category I or II and are in good physical health as judged by a thorough history and physical examination;
6. Patients without infections in the area of the impacted teeth;
7. Patients must agree to refrain from ingesting any systemic or applying any topical analgesic medication for 3 days or 5 half-lives of the drug prior to and during the study;
8. No alcohol for a minimum of 24 hours prior to the surgery;
9. Female patients must be of non-child bearing potential, defined as postmenopausal for more than 1 year or surgically sterile (hysterectomy, tubal ligation/occlusion) or practicing an acceptable method of contraception (hormonal oral, patch, or implant, double barrier method, intrauterine device, vasectomized or same sex partner, or abstinence). Patients using hormonal birth control must have been on a stable dose of treatment for at least 30 days and received at least 1 cycle of treatment prior to randomization. At Screening and at the day of surgery, all females of childbearing potential must have a negative (serum at screening and urine on day of surgery 1) pregnancy test and not be breastfeeding;
10. Patients must have a negative urine drug screen for drugs of abuse at Screening and on the day of surgery. At the discretion of the Principal Investigator, a positive drug screen result may be permitted if the patient has been on a stable dose of an allowed medication for >30 days;
11. Patients who are scheduled to undergo the surgical removal of up to 4 third molars of which at least two have to be mandibular molars with a difficulty rating of 4 or 5 and meeting the following criteria:

    * two full bony impactions
    * two partial bony impactions
    * one full bony impaction in combination with one partial bony impaction (see Appendix 1 for Impaction Difficulty Rating Scale);
12. Patients able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon the research site's judgment.

Exclusion Criteria:

1. Patients with a history of any significant medical condition that, in the opinion of the Principal Investigator or his designee, would place the patient at increased risk such as: hepatic, renal, endocrine, cardiac, neurological, psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorders, including glaucoma, diabetes, emphysema, and chronic bronchitis;
2. Patients with a history of any type of malignancy within the past 5 years other than minor skin related cancers;
3. Patients with a history of alcohol or substance abuse in the past three years according to Diagnostic and Statistical Manual (DSM) V and who do not satisfy Inclusion Criteria 10 (including a positive urine drug screen test);
4. Patients with a known allergy or hypersensitivity to any local anesthetic drug, acetaminophen, ibuprofen, or other NSAIDS;
5. Patients who are taking any concomitant medications that might confound assessments of pain relief, such as psychotropic drugs, antidepressants, sedative hypnotics or any analgesics taken within three days or five times of their elimination half-lives, whichever is longer. Selective serotonin reuptake inhibitors (SSRIs) and selective noradrenaline reuptake inhibitors (SNRIs) are permitted if the patient has been on a stable dose for at least 30 days prior to screening;
6. Patients who have smoked or chewed tobacco-containing substances within 48 hours prior to the day of surgery;
7. Patients judged by the Principal Investigator to be unable or unwilling to comply with the requirements of the protocol;
8. Patients who have used an investigational drug within 30 days prior to the screening day or have previously participated in any Nevakar trial;
9. Patients who have donated blood within 3 months prior to the screening day;
10. Patients who are employees or relatives of employees of JBR Clinical Research or Nevakar, Inc.
11. Patients with liver function tests (ALT, AST) that are above the normal reference range.

    -

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lang, MD, Study Director — Nevakar, Inc.
Locations (1):
- JBR, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from April 2019 till July 2019 from the site
Pre-assignment Details: A total of 226 participants were screened from Day-30 to Day 0 before getting randomized
Groups:
- High Dose APAP: Acetaminophen (APAP) administered post-operatively at a high dose
- Low Dose APAP: Acetaminophen (APAP) administered post-operatively at a low dose
- Placebo: Placebo given post-operatively
Period: Overall Study
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Started | 44 | 44 | 22
Completed | 43 | 44 | 21
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was the Safety Population that included all randomized participants who received the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose APAP | Low Dose APAP | Placebo | Total
Number analyzed (Participants) | 44 | 44 | 22 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.7 (2.06) | 18.8 (2.31) | 19.3 (2.42) | 18.9 (2.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 11 | 58
  Male | 19 | 22 | 11 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race-Asian | 1 | 0 | 0 | 1
  Race-White | 39 | 39 | 22 | 100
  Race-Others | 2 | 4 | 0 | 6
  Race-Black or African American | 1 | 0 | 0 | 1
  Race- Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Ethnicity-Hispanic or Latino | 9 | 8 | 1 | 18
  Ethinicity-Not Hispanic or Latino | 35 | 36 | 21 | 92
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.45 (4.124) | 24.33 (3.762) | 25.49 (4.869) | 24.61 (4.130)
Categorical pain intensity score [Count of Participants; unit: Participants]
  None (0) | 0 | 0 | 0 | 0
  Mild (1) | 0 | 0 | 0 | 0
  Moderate (2) | 14 | 11 | 10 | 35
  Severe (3) | 30 | 33 | 12 | 75
NRS pain intensity [Count of Participants; unit: Participants]
  0 = No pain | 0 | 0 | 0 | 0
  1 | 0 | 0 | 0 | 0
  2 | 0 | 0 | 0 | 0
  3 | 0 | 0 | 0 | 0
  4 | 0 | 0 | 0 | 0
  5 | 1 | 1 | 1 | 3
  6 | 11 | 7 | 8 | 26
  7 | 13 | 12 | 6 | 31
  8 | 13 | 18 | 7 | 38
  9 | 3 | 5 | 0 | 8
  10 = Worst imaginable pain | 3 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference From 0 to 24 Hours (SPID24) Based on the 11 Point Numeric Pain Rating Scale
Description: Pain Intensity was self-reported over 24 hours, using a pain rating of 0-10 on the Numerical Rating Scale (NRS), with score between 0-10 (0= no pain; 10 = worst imaginable pain). Time weighted sum of pain intensity difference from 0 to 24 hours was reported. Pain Intensity (PI-NPRS) was collected at initiation of Dose 1 (T0) and post dose 0.5, 0.75, 1, 1.25, 1.75, 2.25 3.25, 4.25, 5.25, 6.25, 7.25, 8.25, 9.25, 10.25, 11.25, 12.25 (± 5 min) and 14.25, 16.25, 18.25, 20.25, 22.25, and 24.25 (± 10 min). SPID24 was include all nominal timepoints from T0 to T24.25 hours. SPID is calculated as Σ[T(i) -T(i-1)] x [(PID(i-1) + PID(i))/2], where T(0)=0, T(i) is the scheduled time, and PID(i) is the pain intensity difference (PID) score at time i. Pain intensity differences were calculated with respect to Baseline. A baseline assessment is defined as the last non-missing result prior to administration of the first dose of study medication.
Time Frame: Baseline (0.0) and 0.5, 0.75, 1, 1.25, 1.75, 2.25 3.25, 4.25, 5.25, 6.25, 7.25, 8.25, 9.25, 10.25, 11.25, 12.25 (± 5 min) and 14.25, 16.25, 18.25, 20.25, 22.25, and 24.25 (± 10 min) hours
Population: The Evaluable Population included all randomized participants who, as documented prior to the breaking of the study blind: (1) met all the inclusion and exclusion criteria and; (2) were administered Dose 1.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 22
score on a scale | -96.80 (6.369) | -100.69 (6.333) | -74.96 (9.055)
Statistical Analysis 1: Comparison: High Dose APAP vs Placebo; Test type: Superiority; p = 0.0258, ANCOVA; LS Mean Difference = -21.84, 90% CI 1-sided [upper limit -7.53], Standard Error of Mean 11.091 — SPID24 was analyzed using ANCOVA model with treatment group as a fixed effect and baseline (BL) Pain Intensity-Numerical Pain Relief Scale (PI-NPRS) as a covariate. The lower limit of one-sided 90% confidence interval (CI) was -∞
Statistical Analysis 2: Comparison: Low Dose APAP vs Placebo; Test type: Superiority; p = 0.0115, ANCOVA; LS Mean Difference = -25.74, 90% CI 1-sided [upper limit -11.35], Standard Error of Mean 11.154 — SPID24 was analyzed using an analysis of covariance (ANCOVA) model with treatment group as a fixed effect and baseline PI-NPRS as a covariate. The lower limit of one-sided 90% CI was -∞

2. Primary Outcome: Sum of Pain Relief From 0 to 24 Hours (TOTPAR24) Based on a 5-point Likert Scale.
Description: Pain Relief Rating (PR) was scored on a 5-point scale (0=no-, 1=a little-, 2=some-, 3=a lot of-, and 4=complete- PR). PR was collected at initiation of Dose 1 (T0) and post dose 0.5, 0.75, 1, 1.25, 1.75, 2.25 3.25, 4.25, 5.25, 6.25, 7.25, 8.25, 9.25, 10.25, 11.25, 12.25 (± 5 min) and 14.25, 16.25, 18.25, 20.25, 22.25, and 24.25 (± 10 min) hours. TOTPAR24 is calculated as Sum ([T(i) - T(i-1)] x (PR(i-1) + PR(i)) / 2), where T(0)=0, T(i) is the actual time, and PR(i) is the pain relief score at time i. and calculated as Σ[T(i) -T(i-1)] x [(PR(i-1) + PR(i))/2], where T(0)=0, T(i) is the scheduled time, and PR(i) is the pain relief (PR) score at time i.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 22
score on a scale | 55.82 (3.024) | 55.24 (3.007) | 43.11 (4.300)
Statistical Analysis 1: Comparison: High Dose APAP vs Placebo; Test type: Superiority; p = 0.0087, ANCOVA; LS Mean Difference = 12.72, 90% CI 1-sided [lower limit 5.92], Standard Error of Mean 5.267 — TOTPAR24 was analyzed using an ANCOVA model with treatment group as a fixed effect and baseline PI-NPRS as a covariate. The upper limit of one-sided 90% CI was +∞
Statistical Analysis 2: Comparison: Low Dose APAP vs Placebo; Test type: Superiority; p = 0.0120, ANCOVA; LS Mean Difference = 12.14, 90% CI 1-sided [lower limit 5.31], Standard Error of Mean 5.297 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Time to Perceptible Pain Relief Confirmed (FPR-C) After Dose 1 Administration Stratified by Baseline Pain Score of Moderate or Severe for the 3 Treatment Groups
Description: Upon initiation of the infusion of Dose 1, the participants were given stopwatch #1 and asked to press the stopwatch when they first perceived any pain relief (first perceptible pain relief [FPR]) ; a record of the time was noted in the participant record.
  If a participant does not record perceptible pain relief and prematurely discontinued from the study prior to 24 hours, then the participant was censored at time of drop out. If a participant does not record perceptible pain relief prior to taking rescue medication, the participant was censored at 24 hours
Time Frame: 0 to 24 Hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 21
hours
  Median time to FPR-C (hours)- for moderate baseline categorical pain intensity score: number analyzed (Participants) | 14 | 11 | 9
  Median time to FPR-C (hours)- for moderate baseline categorical pain intensity score | 0.215 [0.080 to 1.000] | 0.160 [0.030 to 0.430] | 0.595 [0.060 to 24.00]
  Median time to FPR-C (hours)- for severe baseline categorical pain intensity score: number analyzed (Participants) | 29 | 33 | 12
  Median time to FPR-C (hours)- for severe baseline categorical pain intensity score | 0.160 [0.030 to 24.00] | 0.220 [0.060 to 24.00] | 0.890 [0.040 to 24.00]

4. Secondary Outcome: Time to Meaningful Perceptible Relief (MPR) Measure Stratified by Baseline Pain Score of Moderate or Severe for the 3 Treatment Groups
Description: Upon initiation of the infusion of Dose 1, the participants were given a second stopwatch and asked to press the stopwatch if and when they feel any meaningful perceptible relief; a record of the time was noted in the participant record.
  If a participant does not record perceptible pain relief and was prematurely discontinued from the study prior to 24 hours, then the participant was censored at time of drop out. If a participant does not record perceptible pain relief prior to taking rescue medication, the participant was censored at 24 hours.
Time Frame: 0 to 24 Hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 21
hours
  Median time to MPR (hours)- for moderate baseline categorical pain intensity score: number analyzed (Participants) | 14 | 11 | 9
  Median time to MPR (hours)- for moderate baseline categorical pain intensity score | 0.660 [0.250 to 24.00] | 0.310 [0.110 to 24.00] | NA [NA to NA] — Median was not estimable as less than 50% of the participants obtained Meaningful Perceptible Relief by 24 hours
  Median time to MPR (hours)- for severe baseline categorical pain intensity score: number analyzed (Participants) | 29 | 33 | 12
  Median time to MPR (hours)- for severe baseline categorical pain intensity score | 0.680 [0.120 to 24.00] | 0.870 [0.150 to 24.00] | NA [NA to NA] — Median was not estimable as less than 50% of the participants obtained Meaningful Perceptible Relief by 24 hours

5. Secondary Outcome: Patient Global Evaluation of the Study Medication
Description: Patients Global Evaluation was assessed on a scale of 0 (Poor), 1 (Fair), 2 (Good), 3 (Very Good) and 4 (Excellent) at 24.25 hours post-dose 1 or at participant withdrawal (if applicable), whichever occurred first. Least squares mean of the score are reported.
Time Frame: 0 to 24 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 42 | 44 | 21
score on a scale | 2.8 (0.16) | 2.7 (0.15) | 2.3 (0.22)

6. Secondary Outcome: Pain Intensity Difference Rating (PID) at Different Timepoints After Dose 1 Administration
Description: Pain Intensity was self-reported over 24 hours, using a pain rating of 0-10 on the Numerical Rating Scale (NRS), with score between 0-10 (0= no pain; 10 = worst imaginable pain). Pain intensity differences were calculated with respect to Baseline at each time point after Dose 1 administration. A baseline assessment was defined as the last non-missing result prior to administration of the first dose of study medication
Time Frame: Baseline (0.0) and 0.5, 0.75, 1, 1.25, 1.75, 2.25 3.25, 4.25, 5.25, 6.25, 7.25, 8.25, 9.25, 10.25, 11.25, 12.25 (± 5 min) and 14.25, 16.25, 18.25, 20.25, 22.25, and 24.25 hours (± 10 min)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 22
score on a scale
  0.5 | -2.5 (1.65) | -3.1 (2.01) | -0.7 (1.28)
  0.75 | -3.3 (1.88) | -3.5 (2.10) | -0.8 (1.40)
  1 | -3.7 (1.89) | -3.8 (2.12) | -0.8 (1.44)
  1.25 | -3.9 (2.02) | -4.0 (2.29) | -0.7 (1.52)
  1.75 | -3.9 (1.97) | -3.7 (2.45) | -0.7 (1.59)
  2.25 | -3.8 (2.16) | -3.6 (2.44) | -0.7 (1.67)
  3.25 | -3.4 (2.32) | -3.0 (2.39) | -0.9 (1.95)
  4.25 | -3.4 (2.40) | -2.9 (2.32) | -0.9 (1.97)
  5.25 | -3.3 (2.48) | -2.8 (2.39) | -2.4 (2.59)
  6.25 | -3.2 (2.48) | -3.5 (2.49) | -3.7 (2.32)
  7.25 | -3.0 (2.61) | -4.1 (2.34) | -4.2 (1.99)
  8.25 | -3.8 (2.72) | -4.4 (2.29) | -3.7 (2.36)
  9.25 | -4.5 (2.89) | -4.7 (2.18) | -3.6 (2.26)
  10.25 | -4.6 (2.71) | -5.0 (1.98) | -3.4 (2.22)
  11.25 | -4.7 (2.44) | -4.5 (1.99) | -3.3 (2.28)
  12.25 | -4.9 (1.85) | -4.5 (2.31) | -2.7 (2.27)
  14.25 | -3.7 (2.13) | -5.0 (2.42) | -2.9 (1.97)
  16.25 | -3.5 (2.29) | -4.4 (2.08) | -2.9 (1.97)
  18.25 | -4.4 (2.34) | -4.5 (2.27) | -3.5 (1.97)
  20.25 | -4.7 (2.04) | -4.9 (2.37) | -3.6 (2.24)
  22.25 | -4.7 (2.25) | -5.0 (2.35) | -3.9 (2.19)
  24.25 | -4.6 (2.29) | -5.1 (2.42) | -4.3 (1.86)

7. Secondary Outcome: Pain Intensity Rating at Different Timepoints After Dose 1 Administration
Description: Pain intensity is reported using the 11-point Numerical Rating Scale (NRS), with score between 0-10 (0= no pain; 10 = worst imaginable pain).
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 22
score on a scale
  0.5 | 4.8 (1.83) | 4.4 (1.97) | 6.1 (1.42)
  0.75 | 4.0 (2.12) | 4.0 (1.98) | 6.0 (1.70)
  1 | 3.6 (1.98) | 3.7 (2.01) | 6.0 (1.68)
  1.25 | 3.4 (2.16) | 3.5 (2.14) | 6.2 (1.89)
  1.75 | 3.5 (2.24) | 3.8 (2.33) | 6.2 (1.94)
  2.25 | 3.6 (2.40) | 3.9 (2.39) | 6.2 (1.97)
  3.25 | 3.9 (2.53) | 4.5 (2.48) | 6.0 (2.17)
  4.25 | 4.0 (2.58) | 4.6 (2.33) | 6.0 (2.21)
  5.25 | 4.0 (2.48) | 4.7 (2.44) | 4.5 (2.56)
  6.25 | 4.2 (2.52) | 4.0 (2.59) | 3.2 (2.11)
  7.25 | 4.3 (2.46) | 3.4 (2.22) | 2.7 (1.86)
  8.25 | 3.5 (2.58) | 3.1 (2.20) | 3.2 (2.30)
  9.25 | 2.9 (2.71) | 2.8 (1.95) | 3.3 (2.25)
  10.25 | 2.8 (2.48) | 2.5 (1.68) | 3.5 (2.15)
  11.25 | 2.7 (2.27) | 3.0 (1.66) | 3.5 (2.24)
  12.25 | 2.5 (1.83) | 3.0 (2.09) | 4.1 (2.32)
  14.25 | 3.6 (2.29) | 2.5 (2.11) | 4.0 (2.08)
  16.25 | 3.8 (2.55) | 3.1 (2.01) | 4.0 (2.21)
  18.25 | 2.9 (2.58) | 3.0 (2.23) | 3.4 (1.99)
  20.25 | 2.7 (2.28) | 2.6 (2.14) | 3.2 (2.22)
  22.25 | 2.6 (2.58) | 2.5 (1.96) | 3.0 (2.16)
  24.25 | 2.8 (2.38) | 2.4 (2.06) | 2.61 (1.71)

8. Secondary Outcome: Pain Relief (PR) Ratings at Each Observation Time After Dose 1 Administration
Description: Pain Relief is reported on a 5-Point Categorical Pain Relief Assessment scale: 0 = No Pain Relief, 1 = A Little Pain Relief, 2 = Some Pain Relief, 3 = A Lot of Pain Relief, 4 = Complete Pain Relief.
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 22
score on a scale
  0.5 | 1.7 (0.95) | 1.8 (0.94) | 0.6 (0.85)
  0.75 | 2.0 (1.02) | 2.0 (0.98) | 0.6 (0.85)
  1 | 2.1 (0.93) | 2.2 (0.96) | 0.6 (0.85)
  1.25 | 2.3 (0.97) | 2.2 (0.99) | 0.6 (0.85)
  1.75 | 2.3 (0.97) | 2.0 (1.07) | 0.6 (0.90)
  2.25 | 2.2 (1.09) | 2.0 (1.05) | 0.6 (0.90)
  3.25 | 2.0 (1.18) | 1.7 (1.12) | 0.8 (1.15)
  4.25 | 2.0 (1.21) | 1.6 (1.12) | 0.7 (1.08)
  5.25 | 1.9 (1.20) | 1.5 (1.21) | 1.5 (1.44)
  6.25 | 1.9 (1.23) | 1.9 (1.15) | 2.1 (1.25)
  7.25 | 1.8 (1.21) | 2.2 (1.03) | 2.5 (1.10)
  8.25 | 2.2 (1.15) | 2.4 (1.06) | 2.2 (1.27)
  9.25 | 2.6 (1.22) | 2.5 (0.93) | 2.1 (1.19)
  10.25 | 2.6 (1.10) | 2.7 (0.80) | 2.0 (1.20)
  11.25 | 2.7 (0.97) | 2.5 (0.87) | 2.0 (1.31)
  12.25 | 2.7 (0.83) | 2.4 (1.04) | 1.6 (1.33)
  14.25 | 2.1 (1.00) | 2.6 (1.04) | 1.8 (1.11)
  16.25 | 2.1 (1.14) | 2.3 (1.06) | 1.8 (1.14)
  18.25 | 2.5 (1.10) | 2.4 (1.02) | 2.1 (1.17)
  20.25 | 2.7 (1.00) | 2.6 (0.95) | 2.2 (1.18)
  22.25 | 2.7 (1.11) | 2.6 (0.94) | 2.3 (1.09)
  24.25 | 2.5 (1.12) | 2.7 (0.99) | 2.5 (0.91)

9. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as time to first dose of rescue medication after Dose 1 or withdrawal from the study for any reason. If a participant does not take rescue medication or withdraw from the study prior to 24 hours, the participant was censored at 24 hours
Time Frame: 0 to 24 Hours
Population: The Evaluable Population included all randomized participant who, as documented prior to the breaking of the study blind: (1) met all the inclusion and exclusion criteria and; (2) were administered Dose 1.
Measure: Median (Full Range); unit: hours
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 21
hours
  Median time to treatment failure- for moderate baseline categorical pain intensity score: number analyzed (Participants) | 14 | 11 | 9
  Median time to treatment failure- for moderate baseline categorical pain intensity score | NA [NA to NA] — Median was not estimable as less than 50% of the participants had treatment failure by 24 hours | NA [NA to NA] — Median was not estimable as less than 50% of the participants had treatment failure by 24 hours | 3.680 [1.100 to 24.00]
  Median time to treatment failure for severe baseline categorical pain intensity score: number analyzed (Participants) | 29 | 33 | 12
  Median time to treatment failure for severe baseline categorical pain intensity score | NA [NA to NA] — Median was not estimable as less than 50% of the participants had treatment failure by 24 hours | NA [NA to NA] — Median was not estimable as less than 50% of the participants had treatment failure by 24 hours | 1.335 [1.030 to 24.00]

10. Other Pre Specified Outcome: Mean Change From Baseline to 24 Hours in Vital Signs (Systolic Blood Pressure)
Description: Change from Baseline in systolic blood pressure is the value at 24 hours minus value at Baseline. Baseline was defined as the last non-missing result prior to administration of the first dose of study drug. Systolic blood pressure is obtained at screening, prior to surgery and at Hours 4, 8, 12, 16, 20 and 24 following initiation of dose (±10 min).
Time Frame: 0 to 24 hours
Population: The Safety Population included all randomized participants who received the study medication. This population was used for all safety summaries.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 21
mm Hg | 1.6 (10.78) | 1.0 (11.39) | 9.2 (10.99)

11. Other Pre Specified Outcome: Mean Change From Baseline to 24 Hours in Vital Signs (Diastolic Blood Pressure)
Description: Change from Baseline in diastolic blood pressure is the value at 24 hours minus value at Baseline. Baseline was defined as the last non-missing result prior to administration of the first dose of study drug. Diastolic blood pressure is obtained at screening, prior to surgery and at Hours 4, 8, 12, 16, 20 and 24 following initiation of dose (±10 min)
Time Frame: 0 to 24 hours
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 21
mm Hg | -0.2 (8.82) | 2.3 (9.56) | 5.2 (11.08)

12. Other Pre Specified Outcome: Mean Change From Baseline to 24 Hours in Vital Signs (Temperature)
Description: Change from Baseline in temperature is the value at 24 hours minus value at Baseline. Baseline was defined as the last non-missing result prior to administration of the first dose of study drug. Temperature is obtained at screening, prior to surgery and at Hours 4, 8, 12, 16, 20 and 24 following initiation of dose (±10 min)
Time Frame: 0 to 24 hours
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 21
degrees Celsius | 0.12 (0.336) | 0.21 (0.275) | 0.06 (0.347)

13. Other Pre Specified Outcome: Mean Change From Baseline to 24 Hours in Vital Signs (Pulse Rate)
Description: Change from Baseline in pulse rate is the value at 24 hours minus value at Baseline. Baseline was defined as the last non-missing result prior to administration of the first dose of study drug. Pulse rate is obtained at screening, prior to surgery and at Hours 4, 8, 12, 16, 20 and 24 following initiation of dose (±10 min)
Time Frame: 0 to 24 hours
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 44 | 21
beats/minute | 5.0 (11.85) | 4.2 (11.58) | 5.7 (11.17)

14. Other Pre Specified Outcome: Mean Change From Baseline to 24 Hours in Vital Signs (Respiratory Rate)
Description: Change from Baseline in respiratory rate was the value at 24 hours minus value at Baseline. Baseline was defined as the last non-missing result prior to administration of the first dose of study drug. Respiratory rate was obtained at screening, prior to surgery and at Hours 4, 8, 12, 16, 20 and 24 following initiation of dose (±10 min)
Time Frame: 0 to 24 hours
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
Number analyzed (Participants) | 43 | 43 | 21
breaths/minute | 0.3 (3.39) | -0.6 (4.12) | -1.3 (3.68)

15. Other Pre Specified Outcome: Area Under the Plasma Concentration-Time Curve From Time of Administration to 24 Hours After Dosing (AUC 0-24h)
Description: The Area Under the Plasma Concentration-Time Curve (AUC) is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption. The values for pharmacokinetic (PK) evaluable population-excluding participants with positive pre-dose concentrations have been populated. The samples were collected at 5 min prior to Dose 1, and at 0.25, 0.5, 0.75, 1.0, 2.0, 4.0, 6.25, 8.0, 8.25, 8.25, 12.0, 12.25, 16.0, 16.25, 18.0, 18.25, 24.25 hours post-dose 1.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1.0, 2.0, 4.0, 6.25, 8.0, 8.25, 8.25, 12.0, 12.25, 16.0, 16.25, 18.0, 18.25, 24.25 hours post-dose
Population: The PK Evaluable Population included all randomized participants who, as documented prior to the breaking of the study blind: (1) met all the inclusion and exclusion criteria and; (2) were administered Dose 1 resulting in an adequate number of quantifiable concentrations to calculate PK parameters.
Measure: Least Squares Mean (Standard Error); unit: microgram*hour/milliliter
Arm/Group | High Dose APAP | Low Dose APAP
Number analyzed (Participants) | 31 | 38
microgram*hour/milliliter | 236326.3081 (1.06026) | 231104.0073 (1.05427)

16. Other Pre Specified Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity])
Description: The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time. The samples were collected at 5 min prior to Dose 1, and at 0.25, 0.5, 0.75, 1.0, 2.0, 4.0, 6.25, 8.0, 8.25, 8.25, 12.0, 12.25, 16.0, 16.25, 18.0, 18.25, 24.25 hours post-dose 1.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter
Arm/Group | High Dose APAP | Low Dose APAP
Number analyzed (Participants) | 42 | 43
hour*nanogram per milliliter | 75925.2553 (22.405) | 55018.1382 (27.089)

17. Other Pre Specified Outcome: Half-life
Description: The half-life (t 1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | High Dose APAP | Low Dose APAP
Number analyzed (Participants) | 42 | 43
hours | 2.565 (0.5774) | 2.360 (0.4134)

18. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The Plasma Concentration (Cmax) is defined as maximum observed concentration
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ml)
Arm/Group | High Dose APAP | Low Dose APAP
Number analyzed (Participants) | 31 | 39
nanogram per milliliter (ng/ml) | 39531.4 (26) | 28495.6 (30)

ADVERSE EVENTS:
Time Frame: Up to 7 days (± 2 days)
Description: An adverse event (AE) is defined as any untoward medical occurrence and does not necessarily have to have causal relationship with the study medication. An AE can therefore be an unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease, which is a change from baseline and is temporally associated with the use of the study medication, whether or not it is considered related to the study medication.
Arm/Group | High Dose APAP | Low Dose APAP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/22
Other Adverse Events (participants affected / at risk) | 9/44 | 13/44 | 7/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose APAP (N=44) | Low Dose APAP (N=44) | Placebo (N=22)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 7 (7) | 8 (8) | 6 (6)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT04018612/Prot_SAP_002.pdf